CLINICAL TRIAL: NCT03882008
Title: Phase IV Open-Label Study to Evaluate Biomarkers to Predict the Efficacy of Abatacept in Subjects With Rheumatoid Arthritis
Brief Title: A Study to Evaluate Biomarkers to Predict Efficacy of Abatacept in Rheumatoid Arthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Kwanghoon (Bobby) Han, Assistant Professor, School of Medicine: Department of Medicine: Rheumatology, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY00004744
Record Dates: First submitted 2018-11-07; First posted 2019-03-20 (Actual); Results first posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Abatacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Abatacept (Experimental): Abatacept 125mg subcutaneous injection weekly for 24 weeks
  Interventions: Drug: Abatacept

INTERVENTIONS:
Drug: Abatacept — All the subjects will receive Abatacept subcutaneous injection once a week for 24 weeks
  Other Names: Orencia

SUMMARY:
The primary objective of this study is to evaluate if baseline levels of T cell associated biomarkers predict efficacy of abatacept during 24 weeks of treatment in patients with moderate to severe active Rheumatoid Arthritis (RA) who have had an inadequate response to conventional disease modifying anti-rheumatic drugs (cDMARDs)

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant, non-nursing female
* Age 18 years or greater
* Body weight less than or equal to 120 kg
* Classification of Rheumatoid Arthritis according to the 1987 ACR criteria or 2010 ACR/EULAR criteria
* Symptoms of Rheumatoid Arthritis present for at least 3 months and less that 10 years prior to Screening.
* Clinical Disease Activity Index (CDAI) greater than or equal to 16, corresponding to moderate to severe disease activity.
* Patients taking oral DMARDs must be on stable doses of DMARDs for at least 4 weeks prior to Abatacept initiation
* Treatment within the past year with either methotrexate, leflunomide, hydroxychloroquine and/or sulfasalazine for greater than or equal to 8 weeks.
* Patients who have received one prior Tumor necrosis factor (TNF) inhibitor must have discontinued etanercept, infliximab, adalimumab, certolizumab, or golimumab for at least 6 months prior to screening.
* Patients taking oral corticosteroids, the dose must be less than or equal to 5mg per day (prednisone or equivalent)
* Females of child bearing potential and males with female partners of child bearing potential may participate in this study only if using a reliable means of contraception

Exclusion Criteria:

* Previous treatment with Abatacept (Orencia)
* Previous treatment with rituximab, tocilizumab, tofacitinib, sarilumab, or anakinra
* Previous treatment with IV immunoglobulin, plasmapheresis, or alkylating agents such as cyclophosphamide
* Intraarticular or parenteral corticosteroids within 4 weeks of screening
* Rheumatic autoimmune disease other than Rheumatoid Arthritis, including Systemic Lupus Erythematosus, primary Sjogren syndrome, spondyloarthritis, systemic sclerosis, dermatomyositis, mixed connective tissue disease, or vasculitis
* Non-rheumatic auto-immune disease including inflammatory bowel disease, psoriasis, multiple sclerosis
* Recurrent or chronic bacterial, viral, fungal, mycobacterial, or other infections including Human immunodeficiency virus (HIV), Hepatitis B, Hepatitis C, latent tuberculosis (TB) (TB not adequately treated)
* Primary or secondary immunodeficiency
* Current, uncontrolled renal, gastrointestinal, endocrine, pulmonary, cardiac, or neurologic disease
* History of malignancy within 10 years prior to screening, except for appropriately treated carcinoma in situ of the cervix or non-melanoma skin carcinoma
* History of alcohol, drug, or chemical abuse within 1 year prior to screening
* Laboratory exclusion criteria at screening including:

  1. estimated glomerular filtration rate (eGFR) <30ml/min
  2. Alanine aminotransferase (ALT) or Aspartate aminotransferase (AST) >1.5 times upper limit of normal
* Major surgery (including joint surgery) within 8 weeks prior to screening or planned major surgery during the study
* Immunization with a live/attenuated vaccine within 4 weeks prior to screening
* Pregnant or nursing women, or women of child bearing potential who plan to become pregnant prior to 14 weeks after the last dose of abatacept treatment
* Patients of reproductive potential not willing to use an effective method of contraception
* Prisoners, or subjects who are compulsory detained

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-05-23 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kwanghoon Han, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Abatacept: Subjects will receive abatacept 125mg subcutaneous injection once a week for 24 doses (24 weeks)
Period: Overall Study
Arm/Group | Abatacept
Started | 25
Completed | 23
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Abatacept
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 18
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With American College of Rheumatology (ACR) 20 Response at Week 14
Description: Baseline levels of T cell-associated biomarkers predict ACR20 response (improvement of 20% in the number of tender and number of swollen joints, and a 20% improvement in three of the following five criteria: patient global assessment, physician global assessment, pain, functional ability measure, erythrocyte sedimentation rate (ESR) or C-reactive protein) with subcutaneous abatacept
Time Frame: 14 Weeks
Measure: Number; unit: participants
Arm/Group | Abatacept
Number analyzed (Participants) | 23
participants | 9

2. Secondary Outcome: Number of Participants With American College of Rheumatology (ACR) 20 Response at Week 24
Description: Baseline levels of T cell associated biomarkers predict ACR20 response (improvement of 20% in the number of tender and number of swollen joints, and a 20% improvement in three of the following five criteria: patient global assessment, physician global assessment, pain, functional ability measure, erythrocyte sedimentation rate (ESR) or C-reactive protein) with subcutaneous abatacept
Time Frame: 24 Weeks
Measure: Number; unit: participants
Arm/Group | Abatacept
Number analyzed (Participants) | 23
participants | 14

3. Secondary Outcome: Number of Participants With American College of Rheumatology (ACR) 50 Response at Week 24
Description: Baseline levels of T cell associated biomarkers predict ACR50 response (improvement of 50% in the number of tender and number of swollen joints, and a 50% improvement in three of the following five criteria: patient global assessment, physician global assessment, pain, functional ability measure, erythrocyte sedimentation rate (ESR) or C-reactive protein) with subcutaneous abatacept
Time Frame: Week 24
Measure: Number; unit: participants
Arm/Group | Abatacept
Number analyzed (Participants) | 23
participants | 10

4. Secondary Outcome: Number of Participants With American College of Rheumatology (ACR) 70 Response at Week 24
Description: Baseline levels of T cell associated biomarkers predict ACR70 response (improvement of 70% in the number of tender and number of swollen joints, and a 70% improvement in three of the following five criteria: patient global assessment, physician global assessment, pain, functional ability measure, erythrocyte sedimentation rate (ESR) or C-reactive protein) with subcutaneous abatacept
Time Frame: Week 24
Measure: Number; unit: participants
Arm/Group | Abatacept
Number analyzed (Participants) | 23
participants | 3

5. Secondary Outcome: Number of Participants With European League Against Rheumatism (EULAR) Good or Moderate Response at Week 24
Description: Baseline levels of T cell associated biomarkers predict EULAR good or moderate response (disease activity index for RA generated from tender and swollen joint count, patient global assessment, ESR or C-reactive protein) with subcutaneous abatacept
Time Frame: Week 24
Measure: Number; unit: participants
Arm/Group | Abatacept
Number analyzed (Participants) | 23
participants | 17

ADVERSE EVENTS:
Time Frame: From time of study drug administration to end of study (week 24 or safety follow-up visit, if needed), up to 39 weeks
Arm/Group | Abatacept
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 8/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Abatacept (N=25)
upper respiratory infection (Infections and infestations) | 3
headaches (Nervous system disorders) | 3
abdominal pain (Gastrointestinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-09): https://cdn.clinicaltrials.gov/large-docs/08/NCT03882008/Prot_SAP_001.pdf